CLINICAL TRIAL: NCT03548714
Title: PT150 (Formerly ORG34517) as a Potential Treatment for Alcohol Dependence-Alcohol Interaction Study
Brief Title: Clinical Trial to Evaluate the Safety of PT150 (Formerly ORG34517) When it is Taken Concurrently With Alcohol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pop Test Oncology LLC (Industry)
Collaborators: Pharmacotherapies for Alcohol and Substance Use Disorders Alliance (Other); Congressionally Directed Medical Research Programs (U.S. Federal Agency); Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Baylor College of Medicine (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AS140026-A3.b; W81XWH-15-2-0077 (Other: RTI International)
Record Dates: First submitted 2018-05-10; First posted 2018-06-07 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Alcohol Dependence; Alcohol Interaction
Keywords: Alcohol; Alcoholic; Alcoholism; Alcohol abuse; Alcohol interaction; Alcohol Use Disorder; Alcohol use; Alcohol dependence; Alcohol dependent; Ethanol abuse; Ethanol use
MeSH Terms: conditions — Alcoholism; Alcohol Drinking | interventions — (11R,13S,17S)-11-(1,3-benzodioxol-5-yl)-17-hydroxy-13-methyl-17-prop-1-ynyl-1,2,6,7,8,11,12,14,15,16-decahydrocyclopenta(a)phenanthren-3-one; Beverages

STUDY DESIGN:
Intervention Model Description: Apart from the Research Pharmacists, all others engaged with this study (participants and study team) will be masked to alcohol challenge order.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PT150 with alcohol consumption (Experimental): Study drug to be administered as a single, fixed dose over a 5-day period. An alcohol challenge (with ethanol or placebo beverage) will be completed on day 1 (pre-treatment), and day-5 (post-treatment), at predetermined times.
  Interventions: Drug: PT150
- PT150 with placebo consumption (Placebo Comparator): Study drug to be administered as a single, fixed dose over a 5-day period. An alcohol challenge (with ethanol or placebo beverage) will be completed on day 1 (pre-treatment), and day-5 (post-treatment), at predetermined times.
  Interventions: Other: Beverage

INTERVENTIONS:
Drug: PT150 — Intervention 1 includes PT150 with alcohol consumption
  Other Names: Formerly ORG34517
  Arms: PT150 with alcohol consumption
Other: Beverage — Alcohol beverage will be prepared by an in-house pharmacist at the MEDVAMC in a volume of 450 ml for a 70 kg individual and adjusted for body weight by varying the volume. Alcohol will be administered in a concentration of 16% alcohol (Everclear, St. Louis, MO) by volume in grape Kool-Aid (Kraft Foods, Northfield, IL). Placebo will be prepared in the same manner but contain 1% alcohol to mask taste.
  Other Names: Placebo drink and ethanol drink
  Arms: PT150 with placebo consumption

SUMMARY:
The purpose of the clinical study is to compare pharmacodynamic and safety endpoints following an alcohol challenge prior to and concurrent with PT150 (study drug) treatment.

DETAILED DESCRIPTION:
This study can be classified as a phase 1, single center, and drug study. This within-subjects experimental procedure will assess the effects of PT150 (900 mg qd) on the subjective effects of alcohol in non-treatment-seeking alcohol-experienced volunteers (to include military service members, veterans and/or civilians). Study duration will be six days; in-house; Day 0 (admission) until day six (final study day and day of discharge). Participants will undergo two alcohol challenges on day 1 separated by 4 hours (one with alcohol, 0.8g/kg; 16% ethanol by volume, and one with placebo beverage, 1% ethanol by volume, randomly ordered) and receive active study drug (PT150) from days 1-5 (after alcohol challenge for day 1). On day 5, the study drug dosing will be followed by two more alcohol challenges (alcohol and placebo beverage randomly ordered). Physiologic (e.g., vital signs, electrocardiogram), subjective and psychometric effects (e.g., mood, urge, craving, stimulant and sedative effects), and breath alcohol levels (BAL) will be obtained after the alcohol challenges. On day six, an electrocardiogram (ECG) will be performed, adverse events (AEs) and symptom checklist will be collected, including symptoms of adrenal insufficiency (AI), and a blood draw for electrolyte levels and cortisol will be collected in the morning followed by breakfast and discharge if laboratory tests are within normal ranges. All serious adverse events will be followed clinically until resolved or clinically stable. Pharmacodynamic and safety endpoints will be assessed during the alcohol challenge prior to, and after 5 days of PT150 treatment, when PT150 has reached steady state. For females, a follow-up visit will be scheduled to occur at least 14 days after the final dose of PT150 is administered to ensure pregnancy does not occur. The objectives of the study are to compare pharmacodynamics and safety endpoints following an alcohol challenge prior to and concurrent with PT150. Given available pre-clinical and clinical evidence for the salutatory effect of glucocorticoid receptor (GR) antagonists on alcohol withdrawal, it was hypothesized that PT150 will not significantly alter pharmacodynamic measures and will be safe and well-tolerated under conditions of alcohol consumption.

ELIGIBILITY:
Inclusion Criteria: - Provide signed and dated informed consent;

* male and female, ages 21 to 64;
* must score <10 on the revised clinical institute withdrawal assessment for alcohol scale (CIWA-Ar) assessed in the context of a blood alcohol level (BAL) ≤ 0.02% to demonstrate that they do not need medical detoxification; must have blood laboratory test results within acceptable limits (normal range as noted per protocol);
* have normal vitals (heart rate 60-100 beats per minute (bpm), systolic blood pressure 90-140 millimeter of mercury (mmHg) and diastolic blood pressure 60-90 mmHg); a baseline electrocardiogram (ECG) that demonstrates clinically normal sinus rhythm, clinically normal conduction, normal QTc, and no clinically significant arrhythmias;
* have a self-reported medical history and brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgement of the admitting physician;
* must be willing to comply with all study procedures and be available for the duration of the study;
* women must either be unable to conceive (i.e., surgically sterilized, sterile, or post-menopausal) or using non-hormonal, medically acceptable contraception during the study and for at least 2 weeks after study completion, with or without additional hormonal contraception Women can be receiving hormone replacement treatment (HRT) as long as the HRT dose has been stable for a period of at least 3 months;
* women must provide negative urine pregnancy tests before study entry (urine), and before alcohol administrations on day 0 or 1 (serum) and on day 5 (urine);
* able to provide proof of age and identity (includes providing full name and date of birth), forms of proof as defined per protocol.

Exclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria for substance use disorders other than alcohol or nicotine or test positive for prescription or illegal substances. With regard to marijuana/tetrahydrocannabinols (THC), an individual must test negative at the baseline. If an individual tests positive they will be given a grace period where they will have the opportunity to return and test negative prior to being enrolled;
* pregnant or nursing;
* receiving HRT where their dose has not been stable for a minimum of 3 months;
* use of concomitant medications (except birth control pills) or other the counter (OTC) supplements for at least 14 days or 5 half-lives (whichever is longer) before the start of the study and for the entire duration of the study. Concomitant medication use includes any prescription, OTC medications, or herbal supplements;
* receiving any non-pharmacotherapy treatments or procedures for which there are precautions for taking concomitantly with PT150 and/or those that interfere with the study;
* have neurological or psychiatric disorders other than Alcohol Use Disorder (AUD);
* history of suicide attempts and/or current suicidal ideation/plan;
* have evidence of untreated or unstable medical illness including: cardiovascular, neuroendocrine, autoimmune, renal, hepatic, or active Human Immucodeficiency Virus (HIV) +, Acquired Immune Deficiency Syndrome (AIDS) infection;
* have a history of medically adverse reactions to alcohol (e.g., loss of consciousness, chest pain, or epileptic seizure) or major alcohol-related medical complications requiring hospitalization (i.e., hepatitis or pancreatitis);
* have contraindication(s) to take the study medications such as renal or hepatic impairment, congenital metabolic disorders, or hypersensitivity to study medication class (i.e., glucosteroid abntagonist);
* have past brain injury/head trauma with current symptoms (e.g., not photophobic, dizziness etc.) or past report of loss of consciousness (LOC) for >30 minutes and/or have been blast-exposed or had LOC >1 minute and current post-concussive symptoms;
* self report more than thirty days' abstinence from alcohol during the three months prior to enrollment/consent;
* current signs or violence or aggression, assessed as part of the consent process;
* a history of adrenal insufficiency or a plasma cortisol level of ≤ 5 microgram per deciliter (mcg/dl) at screening or intake;
* participation in a pharmaceutical trial or exposure to investigational drugs within 1 month of the screening visit;
* currently seeking treatment for AUD
* have any other illness, condition, or use medication (psychotropic or antiretroviral), which in the opinion of the principal investigator (PI) and/or the admitting physician would preclude safe and/or successful completion of the study.
* Have cortisol levels > 5 mcg/dl but < 18 mcg/dL at baseline and an ACTH stimulation test that does not rule out adrenal insufficiency. Those with cortisol levels > 5 mcg/dl but < 18 mcg/dL at baseline and cortisol levels ≥ 18 after stimulation testing can be enrolled.
* Have been treated with any form of corticosteroid in the past 30 days.
* Have a history of endometrial hyperplasia, endometrial cancer, uterine polyps, or unexplained vaginal bleeding.
* Have uncontrolled hypertension (systolic blood pressure >140 mmHg and diastolic blood pressure >90 mmHg).
* Have potassium levels below the normal reference range. Low serum potassium must be corrected prior to dosing in patients with abnormal baseline potassium levels.
* Men taking testosterone replacement therapy.
* Men or women currently interested in fertility.
* Have underlying inflammatory or auto-immune disorders.
* Have elevated thyroid stimulating hormone (TSH) levels.
* Have diabetes.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Change in Breath-alcohol levels (BALs) - Cmax | from post-alcohol challenge pre-treatment (day 1)to post alcohol with concurrent intreatment (day 5)
  Mean estimates of Cmax (observed maximum concentration after alcohol challenge) will be calculated and compared from post-alcohol challenge pre-treatment (day 1) to post alcohol challenge with concurrent treatment (day 5).
Change in Breath-alcohol levels (BALs) - Tmax | from post-alcohol challenge pre-treatment (day 1)to post alcohol with concurrent treatment (day 5)
  Mean estimates of Tmax (time of occurrence of Cmax) will be calculated and compared from post-alcohol challenge pre-treatment (day 1) to post alcohol challenge with concurrent treatment (day 5).
Change in Breath-alcohol levels (BALs) - AUC | from post-alcohol challenge pre-treatment (day 1) to post alcohol with concurrent treatment (day 5)
  Mean estimates of AUC (area under the concentration curve through 2 hours post-alcohol challenge) will be calculated and compared from post-alcohol challenge pre-treatment (day 1) to post alcohol challenge with concurrent treatment (day 5).
Change in blood pressure | from post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
  For each alcohol challenge on Days 1 and 5, the change in blood pressure (systolic and diastolic) is computed as the difference in blood pressure measurements taken during the 2 hours after the alcohol challenges on days 1 and 5 and the ones collected immediately prior to that alcohol challenge. Mean changes are then calculated and compared from both post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
Change in Heart Rate (Pulse) | from post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
  For each alcohol challenge on days 1 and 5, the change in heart rate (pulse) is computed as the difference in heart rate measurements taken during the 2 hours after the alcohol challenges on days 1 and 5 and the ones collected immediately prior to that alcohol challenge. Mean changes are then calculated and compared from both post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5).
Change in ECG abnormalities | from pre-treatment (baseline) to post-treatment (day 6)
  ECG abnormalities (normal, abnormal but not clinically significant, clinically significant abnormal) will be compared between pre-treatment (baseline, day 1 AM) to post-treatment (days 1 through 6)
Change in Positive Affect score from the Positive and Negative Affect Schedule (PANAS) | from post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
  Positive changes in Positive Affect score indicate an increased positive affect. For each alcohol challenge on Days 1 and 5, the change in the positive affect scores are computed as the difference in scores taken during the 2 hours after the alcohol challenges on days 1 and 5 and the ones collected immediately prior to that alcohol challenge. Mean changes are then calculated and compared from both post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
Change in Negative Affect score from the Positive and Negative Affect Schedule (PANAS) | from post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
  Negative changes in Negative Affect score indicate a decreased negative effect post-challenge. For each alcohol challenge on Days 1 and 5, the change in the negative affect scores are computed as the difference in scores taken during the 2 hours after the alcohol challenges on days 1 and 5 and the ones collected immediately prior to that alcohol challenge. Mean changes are then calculated and compared from both post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
Change in Alcohol Urge Questionnaire (AUQ) score | from post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
  The change in AUQ score reflects the participant's thoughts and feelings about drinking, with negative score changes indicating a decrease in craving post-challenge. For each alcohol challenge on Days 1 and 5, the change in the AUQ scores are computed as the difference in scores taken during the 2 hours after the alcohol challenges on days 1 and 5 and the ones collected immediately prior to that alcohol challenge. Mean changes are then calculated and compared from both post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
Change in Biphasic Alcohol Effects Scale (BAES) Sedative effects | from post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
  : The change in BAES sedative effects measures the sedative effects of alcohol, with a positive score change indicating an increase in sedation. For each alcohol challenge on Days 1 and 5, the change in the BAES sedative effects scores are computed as the difference in scores taken during the 2 hours after the alcohol challenges on days 1 and 5 and the ones collected immediately prior to that alcohol challenge. Mean changes are then calculated and compared from both post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
Change in Biphasic Alcohol Effects Scale (BAES) Stimulant effects | from post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
  The change in BAES stimulant effects measures the stimulant effects of alcohol, with a positive score change indicating an increase in stimulation. For each alcohol challenge on Days 1 and 5, the change in the BAES stimulant effects scores are computed as the difference in scores taken during the 2 hours after the alcohol challenges on days 1 and 5 and the ones collected immediately prior to that alcohol challenge. Mean changes are then calculated and compared from both post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
Change in Addiction Research Center Inventory (ARCI) score - Pentobarbital-Chlorpromazine-Alcohol Group Scale | from post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
  The Pentobarbital-Chlorpromazine-Alcohol Group (PCAG) Scale of the ARCI assesses the subjective effects of those psychologically active drugs, with positive score changes indicating an increase in sedation. For each alcohol challenge on Days 1 and 5, the change in the ARCI PCAG scale scores are computed as the difference in scores taken during the 2 hours after the alcohol challenges on days 1 and 5 and the ones collected immediately prior to that alcohol challenge. Mean changes are then calculated and compared from both post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
Change in Addiction Research Center Inventory (ARCI) score - Amphetamine Scale | from post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
  The Amphetamine Scale of the ARCI assesses the subjective effects of that psychologically active drug, with positive score changes indicating an increase in stimulation. For each alcohol challenge on Days 1 and 5, the change in the ARCI amphetamine scale scores are computed as the difference in scores taken during the 2 hours after the alcohol challenges on days 1 and 5 and the ones collected immediately prior to that alcohol challenge. Mean changes are then calculated and compared from both post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
Change in Addiction Research Center Inventory (ARCI) score - Morphine-Benzedrine Group (MBG) Scale | from post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
  The Morphine-Benzedrine Group Scale of the ARCI assesses the subjective effects of those psychologically active drugs, with positive score changes indicating an increase in euphoria/mood elevation. For each alcohol challenge on Days 1 and 5, the change in the ARCI MBG scale scores are computed as the difference in scores taken during the 2 hours after the alcohol challenges on days 1 and 5 and the ones collected immediately prior to that alcohol challenge. Mean changes are then calculated and compared from both post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
Change in Addiction Research Center Inventory (ARCI) score - LSD Scale | from post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
  The LSD Scale of the ARCI assesses the subjective effects of that psychologically active drug, with positive score changes indicating an increase in dysphoric and psychotomimetic changes. For each alcohol challenge on Days 1 and 5, the change in the ARCI LSD scale scores are computed as the difference in scores taken during the 2 hours after the alcohol challenges on days 1 and 5 and the ones collected immediately prior to that alcohol challenge. Mean changes are then calculated and compared from both post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
Change in Addiction Research Center Inventory (ARCI) score - Benzedrine Group Scale | from post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
  The Benzedrine Group Scale of the ARCI assesses the subjective effects of those psychologically active drugs, with positive score changes indicating an increase in intellectual efficiency and energy. For each alcohol challenge on Days 1 and 5, the change in the ARCI Benzedrine scale scores are computed as the difference in scores taken during the 2 hours after the alcohol challenges on days 1 and 5 and the ones collected immediately prior to that alcohol challenge. Mean changes are then calculated and compared from both post-alcohol challenge pre-treatment (day 1) to post-alcohol challenge with concurrent treatment (day 5)
Differences in the adverse events | from pre-treatment (day 1) to post-treatment (day 5)
  Number of adverse events on day 1 (pre-treatment) will be compared to the number of adverse events on Day 5 (post-treatment). Proportion of patients experiencing an adverse event on day 1 (pre-treatment) may also be compared to the proportion of patients experiencing an adverse event on day 5 (post-treatment).

SECONDARY OUTCOMES:
Cognitive Assessment - Hopkins Verbal Learning Task-Revised (HLVT-R) Total Recall Score | from pre-treatment (day 1) to post-treatment (day 5)
  . Change in cognitive effects, measured by the HVLT-R Total Recall scores, will be compared between the day 1 alcohol challenge (pre-treatment) and the day 5 alcohol challenge day 5 (post-treatment).
Cognitive Assessment - Hopkins Verbal Learning Task-Revised (HLVT-R) Delayed Recall Score | from pre-treatment (day 1) to post-treatment (day 5)
  . Change in cognitive effects, measured by the HVLT-R Delayed Recall scores, will be compared between the day 1 alcohol challenge (pre-treatment) and the day 5 alcohol challenge day 5 (post-treatment).
Cognitive Assessment - Hopkins Verbal Learning Task-Revised (HLVT-R) Percent Retained Score | from pre-treatment (day 1) to post-treatment (day 5)
  . Change in cognitive effects, measured by the HVLT-R Percent Retained scores, will be compared between the day 1 alcohol challenge (pre-treatment) and the day 5 alcohol challenge day 5 (post-treatment).
Cognitive Assessment - Hopkins Verbal Learning Task-Revised (HLVT-R) Discrimination Index Score | from pre-treatment (day 1) to post-treatment (day 5)
  . Change in cognitive effects, measured by the HVLT-R Discrimination Index scores, will be compared between the day 1 alcohol challenge (pre-treatment) and the day 5 alcohol challenge day 5 (post-treatment).
Cognitive Assessment - Dual n-Back (DNB) auditory trial accuracy score | from pre-treatment (day 1) to post-treatment (day 5)
  Change in cognitive effects, measured by the DNB auditory trial accuracy scores, will be compared between the day 1 alcohol challenge (pre-treatment) and the day 5 alcohol challenge (post-treatment).
Cognitive Assessment - Dual n-Back (DNB) visual trial accuracy score | from pre-treatment (day 1) to post-treatment (day 5)
  Change in cognitive effects, measured by the DNB visual trial accuracy scores, will be compared between the day 1 alcohol challenge (pre-treatment) and the day 5 alcohol challenge (post-treatment).
Cognitive Assessment - Dual n-Back (DNB) auditory reaction time | from pre-treatment (day 1) to post-treatment (day 5)
  Change in cognitive effects, measured by the DNB auditory reaction times, will be compared between the day 1 alcohol challenge (pre-treatment) and the day 5 alcohol challenge (post-treatment).
Cognitive Assessment - Dual n-Back (DNB) visual reaction time | from pre-treatment (day 1) to post-treatment (day 5)
  Change in cognitive effects, measured by the DNB visual reaction time, will be compared between the day 1 alcohol challenge (pre-treatment) and the day 5 alcohol challenge (post-treatment).
Cognitive Assessment - Continuous Performance Task-2 (CPT) errors of commission score | from pre-treatment (day 1) to post-treatment (day 5)
  Change in cognitive effects, measured by the CPT errors of commission score, will be compared between the day 1 alcohol challenge (pre-treatment) and the day 5 alcohol challenge (post-treatment).
Cognitive Assessment - Continuous Performance Task-2 (CPT) errors of ommission score | from pre-treatment (day 1) to post-treatment (day 5)
  Change in cognitive effects, measured by the CPT errors of ommission score, will be compared between the day 1 alcohol challenge (pre-treatment) and the day 5 alcohol challenge (post-treatment).
Cognitive Assessment - Continuous Performance Task-2 (CPT) errors of perseveration score | from pre-treatment (day 1) to post-treatment (day 5)
  Change in cognitive effects, measured by the CPT errors of perseveration score, will be compared between the day 1 alcohol challenge (pre-treatment) and the day 5 alcohol challenge (post-treatment).
Cognitive Assessment - Continuous Performance Task-2 (CPT) reaction time | from pre-treatment (day 1) to post-treatment (day 5)
  Change in cognitive effects, measured by the CPT reaction time, will be compared between the day 1 alcohol challenge (pre-treatment) and the day 5 alcohol challenge (post-treatment).
Psychomotor Assessment - One Legged Stand (OLS) | from pre-treatment (day 1) to post-treatment (day 5)
  Change in psychomotor effects, measured by the OLS, will be compared between the day 1 alcohol challenge (pre-treatment) and the day 5 alcohol challenge (post-treatment).
Psychomotor Assessment - Walk and Turn (WAT) | from pre-treatment (day 1) to post-treatment (day 5)
  Change in psychomotor effects, measured by the WAT, will be compared between the day 1 alcohol challenge (pre-treatment) and the day 5 alcohol challenge (post-treatment).

CONTACTS AND LOCATIONS:
Locations (1):
- Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with a registry per the data sharing plans of the Consortium.

REFERENCES:
- [Background] Reynolds AR, Saunders MA, Brewton HW, Winchester SR, Elgumati IS, Prendergast MA. Acute oral administration of the novel, competitive and selective glucocorticoid receptor antagonist ORG 34517 reduces the severity of ethanol withdrawal and related hypothalamic-pituitary-adrenal axis activation. Drug Alcohol Depend. 2015 Sep 1;154:100-4. doi: 10.1016/j.drugalcdep.2015.06.018. Epub 2015 Jun 22. PMID 26143299
- [Background] Vendruscolo LF, Estey D, Goodell V, Macshane LG, Logrip ML, Schlosburg JE, McGinn MA, Zamora-Martinez ER, Belanoff JK, Hunt HJ, Sanna PP, George O, Koob GF, Edwards S, Mason BJ. Glucocorticoid receptor antagonism decreases alcohol seeking in alcohol-dependent individuals. J Clin Invest. 2015 Aug 3;125(8):3193-7. doi: 10.1172/JCI79828. Epub 2015 Jun 29. PMID 26121746
- [Derived] Morice C, Baker DG, Patel MM, Nolen TL, Nowak K, Hirsch S, Kosten TR, Verrico CD. A randomized trial of safety and pharmacodynamic interactions between a selective glucocorticoid receptor antagonist, PT150, and ethanol in healthy volunteers. Sci Rep. 2021 May 10;11(1):9876. doi: 10.1038/s41598-021-88609-6. PMID 33972573